| Statistical Analysis Plan |
|---|
| A Phase 2, Randomized, Double-blind, Placebo-Controlled Efficacy, Pharmacokinetics and Safety Study o |
| CA-008 in Subjects Undergoing Total Knee Arthroplasty |

**NCT NUMBER:** 

**OFFICIAL TITLE:** 

NCT03731364

# **DOCUMENT DATE:**

24 April 2019



#### STATISTICAL ANALYSIS PLAN FOR FINAL PILOT STAGE

A Phase 2, Randomized, Double-blind, Placebo-controlled Efficacy, Pharmacokinetics and Safety Study of CA-008 in Subjects Undergoing Total Knee Arthroplasty

**Protocol Number: CA-PS-203** 

Protocol Version 3.2 (19FEB2019)

SPONSORED BY

Concentric Analgesics, Inc.

PREPARED BY
Lotus Clinical Research®, LLC
100 W California Blvd, Unit 25
Pasadena, CA 91105
626-397-2390 office
info@LotusCR.com
www.LotusCR.com

This document is confidential and proprietary to **Concentric Analgesics, Inc.** Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Concentric Analgesics, Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

Statistical Analysis Plan Date: 24APR2019

# **DOCUMENT VERSION CONTROL**

| Version Number | Date | Comments/Changes |
|----------------|-----------|-----------------------------------|
| V1.0 | 13MAR2019 | SAP (Pilot Stage) |
| V2.0 | 24APR2019 | Updated to refer to Protocol v3.2 |


Statistical Analysis Plan
Date: 24APR2019

#### **APPROVALS**

DocuSigned by: Author: Song lion Signer Name: Song Liou Signing Reason: I am the author of this document Signing Time: 4/29/2019 3:37:21 PM PDT 85C80776CFA1404FB9C34B43BB0AA100 29-Apr-19 Song Liou Date: Biostatistician Lotus Clinical Research®, LLC DocuSigned by: nnifer Neyyer Signer Name: Jennifer Nezzer Reviewed: Signing Reason: I have reviewed this document Signing Time: 4/30/2019 1:22:08 PM PDT F51546CD923C410C87CAB1F62D450C79 30-Apr-19 Jennifer Nezzer Date: Director, Biometrics Lotus Clinical Research®, LLC DocuSigned by: Mike Royal Signer Name: Mike Royal Approved: Signing Reason: I approve this document Signing Time: 5/1/2019 7:42:40 AM PDT 608C20EC5FAD4832ADC799E971759505 01-May-19 Mike A. Royal, MD, JD, MBA Date: **Chief Medical Officer** Concentric Analgesics Inc.


Statistical Analysis Plan Date: 24APR2019

# **TABLE OF CONTENTS**

| 1. | PURPOSE OF THE ANALYSES | 9 |
|-------|---------------------------------------------------|------|
| 2. | PROTOCOL SUMMARY | 9 |
| 2.1 | Study Objectives | 9 |
| 2.1.1 | Pilot Stage of the Study | 9 |
| 2.1.2 | Second Stage of the Study | . 10 |
| 2.2 | Overall Study Design and Plan | . 10 |
| 2.2.1 | Study Stopping Rules | . 11 |
| 2.2.2 | Study Population | . 13 |
| 2.2.3 | Treatment Regimens | . 13 |
| 2.2.4 | Treatment Group Assignments or Randomization | . 13 |
| 2.2.5 | Sample Size Determination | . 13 |
| 3. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | . 13 |
| 4. | SUBJECT POPULATIONS | . 15 |
| 4.1 | Analysis Populations | . 15 |
| 4.2 | Disposition of Subjects | . 15 |
| 4.3 | Protocol Deviations | . 16 |
| 5. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | . 16 |
| 5.1 | Demographics and Baseline Characteristics | . 16 |
| 5.2 | Medical/Surgical History | . 16 |
| 5.3 | Prior and Concomitant Medications | . 17 |
| 6. | MEASUREMENTS OF TREATMENT EXPOSURE AND COMPLIANCE | . 17 |
| 7. | EFFICACY EVALUATION | . 18 |
| 7.1 | Handling of Dropouts or Missing Data | . 18 |
| 7.2 | Assessment Time Windows | . 19 |
| 7.3 | Efficacy Endpoints for Pilot Stage | . 19 |
| 7.3.1 | Primary Efficacy Endpoint | . 19 |
| 7.3.2 | Key Secondary Efficacy Endpoints | . 20 |
| 7.4 | Analysis Methods | . 20 |

| 7.4.1 | NRS Measurements | . 20 |
|---|---|---|
| 7.4.2 | Mean Pain Intensity Scores at T96h (Primary Efficacy Endpoint) | . 21 |
| 7.4.3 | AUC 0-96h at Rest (Secondary Efficacy Endpoint) | . 21 |
| 7.4.4 | Opioid Free (OF) 0-96h (Secondary Efficacy Endpoint) | . 22 |
| 7.4.5 | Total Opioid Consumption (OC) in Daily Oral Morphine equivalents 0-96h (Secondary Efficacy Endpoint) | . 22 |
| 8. | SAFETY EVALUATION | . 23 |
| 8.1 | Overview of Safety Analysis Methods | . 23 |
| 8.2 | Adverse Events and SAEs | . 24 |
| 8.3 | Physical Examination | . 26 |
| 8.4 | Vital Signs | . 27 |
| 8.5 | Surgical Site Assessments and Rebound (or Worsening) Pain Assessments | . 27 |
| 8.6 | Neurosensory Test | . 27 |
| 8.7 | X-ray of the Operated Knee | . 27 |
| 8.8 | ECG | . 28 |
| 8.9 | Clinical Laboratory Test Results | . 28 |
| 8.10 | Drugs of Abuse and Alcohol Screens, Pregnancy Test | . 28 |
| 8.11 | Subject pain Assessment Training and Surgery Details | . 28 |
| 9. | PHARMACOKINETIC EVALUATION | . 29 |
| 10. | OTHER ANALYSES | . 29 |
| 11. | INTERIM ANALYSES | . 29 |
| 12. | REFERENCES | . 29 |
| 13. | APPENDICES | . 30 |
| 13.1 | Planned Tables, Figures and Listings | . 30 |
| 13.1.1 | Tables | . 30 |
| 13.1.2 | Listings | . 32 |
| 11 | DOCUMENT HISTORY | 33 |

Statistical Analysis Plan Date: 24APR2019

# **LIST OF IN-TEXT TABLES AND FIGURES**

| Table 2-1 | Protocol-Specified Visits and Visit Windows | 11 |
|-----------|------------------------------------------------------|----|
| Table 2-2 | Study Stopping Rules | 12 |
| Table 3 | Equianalgesic Conversion Table | 23 |
| Table 4 | Table of Imputation Rules for Missing AE Start Dates | 26 |


# LIST OF ABBREVIATIONS (COMMONLY USED)

ADaM Analysis Data Model

ADLs Actives of Daily Living

AE Adverse Event

ANOVA Analysis of variance

ATC Anatomical Therapeutic Chemical

AUC Area Under the Curve

BMI Body Mass Index

CDER Center for Drug Evaluation and Research

CP Completer

CRF Case Report Form

CRO Clinical Research Organization

CSR Clinical Study Report

ECG Electrocardiogram

ET Early Termination

FDA Food and Drug Administration

ICF Informed Consent Form

ICH International Conference on Harmonization

IGE Investigator Global Evaluation

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

MED morphine equivalent dose

NRS Numerical Rating Scale for Pain Intensity

OC Opioid Consumption in morphine equivalent dose

OF Opioid-Free days

PACU Post-Anesthesia Care Unit

PE Physical Examination


PGE Patient Global Evaluation

PK Pharmacokinetic
PT Preferred Term
QOL Quality of Life

SAE Serious Adverse Event/Experience

SAP Statistical Analysis Plan

SD Standard Deviation

SDTM Standard Data Table Model

SOC System Organ Class

SRC Safety Review Committee

TKA Total Knee Arthroplasty

TEAE Treatment Emergent Adverse Event

WHO World Health Organization

WOCF Worst Observation Carried Forward


#### 1. PURPOSE OF THE ANALYSES

Statistical Analysis Plan

Date: 24APR2019

This statistical analysis plan (SAP) is based on protocol number CA-PS-203 Version 3.2 (19FEB2019) from Concentric Analgesics, Inc. This SAP will focus on analyses that will be performed on data collected during the pilot stage of the study. A final SAP was planned to be created and signed off that would provide the full description of the analyses that will be performed for the Pilot Stage and the data collected in Stage 2, however, after enrollment of the 3<sup>rd</sup> Cohort of the Pilot Stage, the sponsor decided to not proceed with Stage 2. Therefore no additional SAP will be created, and no additional analyses are planned.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonization (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials, the most recent ICH E3 Guideline and the Guidance for Industry: Structure and Content of Clinical Study and the most recent FDA draft Guidance for Industry - Analgesic Indications: Developing Drug and Biological Products, dated February 2014.

This SAP describes the data collected during the pilot stage that will be analyzed and the efficacy assessments that will be evaluated for the analysis of Pilot stage. This SAP provides details of the specific statistical methods that will be used for that analysis.

#### 2. PROTOCOL SUMMARY

#### 2.1 Study Objectives

# 2.1.1 Pilot Stage of the Study

# 2.1.1.1 Primary Objective

 To evaluate the efficacy of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective total knee arthroplasty (TKA).

# 2.1.1.2 Secondary Objective

To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective TKA.


 To evaluate the Pharmacokinetic (PK) profile of a single intraoperative administration of CA-008 in subjects undergoing an elective TKA.

To evaluate the opioid-sparing effect of CA-008 vs. placebo.

# 2.1.2 Second Stage of the Study

To be updated in Final SAP.

# 2.2 Overall Study Design and Plan

This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled, parallel design study evaluating, in a pilot stage of the study involving 3 exploratory cohorts, each with a single dose of CA-008 vs. placebo injected/instilled during an elective TKA.

After an interim unblinded analysis of the pilot stage results from Cohort #1, and review of those Cohort 1 topline results (the subject of a previously executed Interim SAP), a protocol amendment was performed to add two additional exploratory cohorts: Cohort #2 CA-008 10 mg vs. placebo and Cohort #3 CA-008 15 mg vs. placebo (with each cohort enrolling n=18 randomized 2:1, respectively) with a volume of 100 mL.

A second stage of the study was anticipated with that second stage using the doses, sample size and number of CA-008 treatment groups vs. placebo to be determined after an interim analysis of the combined cohort #1 - cohort #3 data in this pilot stage. However, after enrollment of Cohort 3 the sponsor decided to end the study after the pilot stage, and Stage 2 will not be performed..

For each subject, the postoperative assessments will be conducted in two parts:

- Inpatient period which continues to 96h (T96h) after completion of study treatment injection (T0).
- Outpatient period which begins on discharge from the inpatient unit through various followup visits to day 29 (D29±2) (W4) after surgery or later if necessary for ongoing safety assessment.

Each subject is expected to be in the study up to 76 days (screening through end of study visit).

The protocol-defined visits are presented in <u>Table 2-1</u>:


Table 2-1 Protocol-Specified Visits and Visit Windows

| Study Phase | Visit Time |
|---------------------------|-------------------------------------------|
| Screening | From days -45 to -1 |
| Prior to Surgery/ Surgery | Day 0 |
| In-Patient (Post Surgery) | Hours 0 (post-surgery), 24, 48, 72 and 96 |
| Follow-up | Days 8(±1 day), 15(±2 days), 29(±2 days) |

Statistical Analysis Plan

Date: 24APR2019

All study assessments are outlined in Table 1 of the Protocol.

# 2.2.1 Study Stopping Rules

Study enrollment will be paused if subjects experience intolerable possibly related TEAEs, as defined:

- 1 or more subjects with any grade 4 "related" TEAE in any of the categories shown in Table 2-2.
- 2 or more subjects with the same grade 3 "related" TEAE in any of the categories shown in Table 2-2.

More details are described in Section 7.3 of the Protocol.

An external independent safety review committee (SRC) will be consulted should a stopping rule be triggered to determine whether it is appropriate to continue with dosing in the study. This committee will be independent of the Sponsor or clinical research organization (CRO) and will in no way be involved with study conduct. The SRC Charter details the membership, roles and responsibilities of the SRC.


Table 2-2 Study Stopping Rules

| Category | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Abnormal Wound Healing: Infection Dehiscence Necrosis | Mild symptoms; clinical or diagnostic observations only; intervention not indicated. No interference with age-appropriate instrumental ADL | Minimal, local or<br>noninvasive<br>intervention<br>indicated; May<br>require local<br>wound care or<br>medical<br>intervention<br>(e.g., dressings<br>or topical<br>medications) | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; limiting ADLs. May require IV antibiotics, antifungals, or antivirals or radiologic intervention. | Life-threatening consequences; urgent intervention indicated |
| ECG/Cardiac<br>issues<br>Vital Signs<br>Labs | Asymptomatic, intervention not indicated | Non-urgent<br>medical<br>intervention<br>indicated | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated | Life-threatening consequences; urgent intervention indicated |
| Focused Neurosensory Testing (performed by trained Investigator) | Mild symptoms | Moderate<br>symptoms;<br>limiting<br>instrumental ADL | Severe<br>symptoms<br>requiring medical<br>intervention;<br>limiting self-care<br>ADL | Life-threatening<br>and urgent<br>intervention<br>indicated |


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

# 2.2.2 Study Population

The study population will consist of adults, aged 18-80 years old inclusive, who are undergoing elective TKA and otherwise meet eligibility criteria (as described in the protocol Sections 8.2.1 and 8.2.2) may be considered for enrollment into the study.

# 2.2.3 Treatment Regimens

Pilot Stage:

Cohort #1: CA-008 5 mg vs. placebo in 100 mL of vehicle

Cohort #2: CA-008 10 mg vs. placebo in 100 mL of vehicle

Cohort #3: CA-008 15 mg vs. placebo in 100 mL of vehicle

## 2.2.4 Treatment Group Assignments or Randomization

In pilot stage of the study, subjects who meet the enrollment criteria will be randomly allocated to receive either an active drug or placebo in a 1:1 (for Cohort #1) or a 2 active: 1 placebo ratio (for Cohorts #2 or #3). This study will use manual randomization.

Subjects who have provided written informed consent will be assigned a unique number in the screening process. This number will be used to identify the subject throughout the study. Once any subject number or randomization number is assigned, it cannot be reassigned to any other subject. Subjects may be rescreened if the screening window is exceeded due to scheduling issues.

# 2.2.5 Sample Size Determination

In the pilot stage, 18 subjects will be randomized to either the active medication or placebo in a 1:1 ratio for Cohort #1. For Cohorts #2 and #3, 18 subjects will be randomized with a ratio of 2 Active: 1 Placebo. Subjects who elect to discontinue study participation after randomization but prior to receiving study treatment will be replaced.

#### 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

This section discusses general policies to be employed in the analysis and reporting of the data from the study. Departures from these general policies may be provided in the specific detailed


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

sections of this SAP. When this situation occurs, the rules set forth in the specific section take precedence over the general policies.

Cohort 1 active and placebo treatments will be presented separately from cohorts 2 and 3 and placebo treatments will not be pooled across all 3 cohorts. Cohort 2 and 3 will have a pooled placebo group and each active dose will be presented separately in summaries and analyses as appropriate.

All continuous study assessments will be summarized by treatment and time point (as applicable) using the descriptive statistics n, mean, SD, median, and range (minimum, and maximum). All of the categorical study assessments will be summarized by treatment and time point (as applicable) using frequency counts and rates of occurrence (%). Changes from baseline for continuous outcomes will be presented as their corresponding continuous measures for post-baseline visits if applicable. All study data will be listed by dose, subject, and time point (as applicable).

No preliminary rounding will be performed; rounding will only occur after the analysis. To round, consider the digit to the right of the last significant digit: if <5, then round down; if ≥5, then round up. Means and medians will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. A percentage of 100% will be reported as 100%. Minimums and maximums will be presented with the same precision as the original data.

All analyses will be performed using the SAS System® version 9.3 or higher. For interim analyses, no SDTM or ADaM data will be generated and data will be analyzed as described in the Interim SAP.

For Final TLFs after Pilot Stage, the domain (Study data tabulation Model [SDTM]) and analysis (Analysis Data Model [ADaM]) data sets will be taken as input to the SAS programs that generate the report-ready tables, figures and listings. The submission ready SDTM and ADaM data sets will be provided to the sponsor along with display deliveries.

The following conventions will be used in the study analysis as needed for interim calculations:

- Time 0 (T0) is the time of completion of study drug administration.
- Time P (TP) is the time of discharge from the post-anesthesia care unit (PACU)


- Day of surgery is defined as Day 0 (D0).
- Assessment visit times are defined by D0 and/or T0.
- Baseline value is defined as the last valid measurement prior to the dosing of study treatment.
- Change from baseline is defined as post-baseline value minus baseline value.
- The date/time of early termination will be the date/time that the subject confirms they no
  longer want to participate in the study, regardless of whether they decide to withdraw from
  all or only some study procedures and regardless of if they return for to the site for
  assessment of wound healing.
- The number of days in the study is computed as: [Date of study completion or withdrawal minus the date of study drug administration] + 1.
- Values that compromise interpretation will not be used in summaries (e.g., values that were obtained post-dose will not be summarized as pre-dose values).

#### 4. SUBJECT POPULATIONS

#### 4.1 Analysis Populations

For the analysis of pilot stage, two analysis populations are defined as follows:

- Safety Population will include all randomized subjects who received any amount of study drug. Subjects will be analyzed by treatment group according to the actual treatment received, i.e., "as treated".
- **PK** Population will include all subjects who receive a full dose of study treatment and complete all PK assessments. Subjects will be analyzed by treatment group according to the actual treatment received, i.e., "as treated".

Analysis population will be determined before the unblinding.

All efficacy and safety analyses will be performed using Safety population for Pilot Stage. PK analyses will be performed using PK population.

#### 4.2 Disposition of Subjects


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

All subjects and the populations for which they qualify will be listed. Subjects who are screened and who fail screening or withdraw consent prior to randomization or are randomized but not treated will be listed and summarized in the disposition summary table. Subjects who are randomized, subject inclusion into each study population, subjects who are treated, subjects who complete follow-up as well as subjects who withdraw early from the study and the reason for withdrawal will be summarized by treatment group and overall in the subject disposition summary table.

#### 4.3 Protocol Deviations

Deviations are categorized as informed consent procedures, inclusion/exclusion criteria, study medication, prohibited medications, study procedures, study drug assignment/treatment, visit or assessment time window, missed visit or assessment and/or other. All protocol deviations will be captured on case report forms (CRFs) and/or documented in site specific logs throughout the study. Deviations will be categorized and classified as major or minor by the project team and the medical monitor after database lock but before unbinding and will be discussed in the CSR. The number of subjects with protocol deviations, both minor and major, will be presented in a data listing and will be summarized by type of deviation and major/minor classification for the ITT population.

#### 5. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

#### 5.1 Demographics and Baseline Characteristics

Demographic variables include age, sex, race, and ethnicity. Baseline characteristics include height (cm), weight (kg), and body mass index (BMI; kg/m²). Demographics and baseline characteristics will be summarized overall and by treatment group using safety population.

# 5.2 Medical/Surgical History

The complete medical and surgical history will include histories of acute, chronic, or infectious disease; surgical or oncologic histories; and any reported conditions affecting major body systems. Subject's medical history will be evaluated by an Investigator for clinical significance. Medical and Surgical history, as collected at screening, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 21.0 to determine system organ class (SOC) and


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

preferred term (PT). Medical histories will be presented in a by-subject listing. Any events that occur prior to the study procedure will be categorized as medical history.

#### 5.3 Prior and Concomitant Medications

Prior medications/therapies are those that stop prior to the start of the study drug administration. Any medication/therapy that stops at or after this time or on going is considered concomitant medication/therapy. Prior and concomitant medications are collected for the 45 days prior to screening and throughout the study. Prior and concomitant medications will be coded using World Health Organization Drug Dictionary Anatomical Therapeutic Chemical (WHO/ATC) classification index version March 1, 2018. The number and percentage of subjects who take concomitant medications will be summarized by drug class and preferred term, overall and by treatment group, for the safety population. All medications and non-medical therapies captured in CRFs will appear in data listings.

#### 6. MEASUREMENTS OF TREATMENT EXPOSURE AND COMPLIANCE

Because study medication is administered as a single dose at the study center by trained study personnel, compliance with respect to study medication will not be calculated. A listing of study drug administration and exposure data will be provided.

After completing the assessments through 96 hours after study medication administration, the diary for at-home use will be distributed to the subject to collect pain intensity (twice daily on NRS) and pain medication through Day 15. Compliance with home diary use will be evaluated based on post-discharge home diary records. Compliance for each subject will be based on the number of days the subject participated in the outpatient study period, defined as:

Where the N of expected NRS records in the diary for each subject is calculated as 2 times the number of days the subject participated in the outpatient portion of the study. The number of days of participation will be calculated as the date of the Day 15 visit or the date of the last study visit (whichever is earlier) minus the date of discharge. NRS recorded prior to a rescue use will not be included in this calculation of compliance. For example, Subject A was discharged on Day 4, if CONFIDENTIAL


Statistical Analysis Plan Protocol Number: CA-PS-203 Date: 24APR2019

this subject discontinues the study on Day 13, then the expected N of NRS records on diary will be 18 (2 \* (13-4)). Assuming Subject A had 10 NRS available from his/her diary, then compliance for this subject would be 55.6% ((10/18) \*100). However, if subject A had discontinued the study on Day 10 (prior to Day 13), then the expected N of NRS for this subject would be 12 (2 \* (10-4)) and compliance would be 83.3% ((10/12) \*100). A summary of compliance will be provided overall and by treatment group. Compliance with recording an NRS prior to rescue in the diary will be calculated as the number of NRS recorded prior to taking rescue medications divided by the number of rescue medication uses recorded.

#### 7. EFFICACY EVALUATION

#### **Handling of Dropouts or Missing Data** 7.1

All efforts will be made to minimize missing data. These efforts will include the following:

- Subjects are required to consent to continuous data collection even after discontinuation of study medication;
- Data collection will continue after subjects take rescue medication.

With the procedures above, it is expected that missing data will be minimal. Missing at random is expected to be a reasonable assumption for this study.

For the endpoints of NRS (at rest and/or after ambulation) in this study, NRS values will be imputed in the following manner:

First, when rescue medication is used, any NRS measured at rest within following window is considered invalid:

- 30 minutes for IV fentanyl
- 2 hours for IV hydromorphone
- 4 hours for PO opioids.

The last NRS prior to the use of any rescue medication will be used to impute subsequent NRS at rest scores for the subsequent protocol-specified time points for measurement of pain intensity through an appropriated time window (as specified above) after the time of the dosing of the rescue medication. Note: if a pre-rescue NRS assessment occurs at the same time as a scheduled assessment, the schedule NRS will be assumed to happen first, and then the pre-

Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

rescue NRS will be assumed to occur. If an NRS assessment occurs at the same time as the time of taking a rescue medication, the NRS will be assumed to be a Pre-rescue medication result. If the NRS time is the same as the end of time window after taking the rescue medication (end of imputation period), then NRS will be considered as occurring before the 4 hours assessment and will be imputed. For example, if a rescue dose (IV morphine) is taken at 1pm, all protocol-scheduled NRS will be imputed with the appropriate NRS value up to and including through 5pm (a 4-hour window). If multiple doses of rescue medication are taken within a 4-hour period, the pre-rescue NRS for the first rescue use will be carried forward continuously until 4 hours past the last use of rescue falling within the continuous window. For example, if rescue is used at Hour 2.3 and Hour 5.1, the pre-rescue NRS at Hour 2.3 will be carried forward till Hour 9.1 (5.1 +4). NRS scores taken after ambulation will be based on reported values and the pre-rescue 4-hour imputation rule will not be used. The scores after ambulation are collected every 12 hours and no ambulation NRS score is collected prior to taking rescue medication.

Intermittent missing pain scores at rest or after ambulation (due to subject sleeping, etc.) will not be imputed, and AUC will be calculated based on non-missing values. For subjects who drop out of the study early, scheduled assessments will first be imputed using the worst prior pain score carried forward (WOCF).

#### 7.2 Assessment Time Windows

For calculations of all AUC endpoints and use of opioid endpoints, the actual <u>dates/times of the assessments</u> will be used in calculations. Thus, while the NRS are intended to be collected at the pre-defined protocol scheduled time points (e.g., Hour 0.5, 1, 2, etc.), it is recognized that operationally the scores are collected as close to the target times as possible but there is some flexibility in terms of the actual times the scores are collected. Thus, to account for this inherent aspect of data collection, the ACTUAL TIMES will be used for the calculation of the AUC. The actual times will be based relative to the time of completion of study drug administration.

Safety assessment summaries will be based on the nominal protocol-specified assessment times.

#### 7.3 Efficacy Endpoints for Pilot Stage

#### 7.3.1 Primary Efficacy Endpoint

Time-specific mean pain intensity scores at T96h for CA-008 vs. placebo.


# 7.3.2 Key Secondary Efficacy Endpoints

Following are key secondary endpoints (in descending order of importance):

- Weighted sum of pain intensity (SPI) assessments = Area Under the Curve (AUC) of the NRS current pain intensity scores from T0 to 96h at rest (AUC<sub>0 to 96h</sub>)
- Percentage of subjects who do not require opioids (i.e., opioid free; OF) from T0 to T96
   (OF<sub>0 to 96h</sub>)
- Total opioid consumption (in daily oral morphine equivalents) from T0 to T96 (OC<sub>0 to 96h</sub>)

# 7.4 Analysis Methods

#### 7.4.1 NRS Measurements

The NRS is an 11-point scale with anchors 0 (no pain) and 10 (worst possible pain). NRS will be assessed as follows:

- During the inpatient stay, NRS at rest beginning with the PACU admission may be assessed once the subject is awake. If the subject is able to provide responses, obtain NRS scores at T0.5, 1, 2, 4, 6, 8, 12, 16, 20, 24, and every 4 hours (if awake at time of assessment) until discharge from the inpatient unit. Time windows: for T0.5 to T2 (±5 min) and from T4 onward (±15 min).
- Pain scores may be skipped between the hours of midnight and 6 a.m., but the subject may not miss two consecutive assessments.
- An additional NRS assessment must be obtained prior to rescue medication request (±15 min). The T12, T24, T48, T72 and T96h assessments must be completed even if the subject is asleep at these times.
- During the inpatient stay, starting on postoperative day 1 (after T24) perform the following each morning at 0800h (±2h) and each evening at 2000h (±2h) document the NRS at rest and after physical therapy or transfers to/from bed or wheelchair (inpatient) or ambulation for approximately 10 yards (inpatient or outpatient). Actual assessment times must be documented. If, however these twice daily assessments coincide with timed assessments of NRS at rest, then the time assessment at rest is used in place of the twice daily


assessments. Resting pain scores are performed on the schedule noted above in the first bullet.

- During the outpatient period (after T96h through W2), instruct the patient to document, if possible, their NRS scores twice daily at 0800h (±4h) and 2000h (±4h) at rest and on ambulation (e.g. with the use of a walker or a cane) for approximately 10 yards. Note that the actual time of these assessments must be documented in the diary whenever possible. Instruct the patient to:
- Obtain the morning NRS assessment prior to taking any pain medication or 2 (±15min) hours after taking any pain medication.
- Obtain the evening NRS assessment 2 (±15min) hours after taking any pain medication.

## 7.4.2 Mean Pain Intensity Scores at T96h (Primary Efficacy Endpoint)

Missing NRS at 96 hours will be handled as discussed in Section 7.1.

Mean NRS scores at 96 hours will be analyzed using a 1-factor (treatment) analysis of variance (ANOVA) model with treatment as the main effect. Descriptive summaries will be presented for each treatment group. Similar ANOVA analyses will also be performed at each time point without imputation for early drop out. In addition, the pain intensity score at Hour 96 and at each time point will be analyzed using Wilcoxon sum-rank test for sensitivity.

#### 7.4.3 AUC 0-96h at Rest (Secondary Efficacy Endpoint)

AUC calculations will be done using the standard trapezoidal rule

$$AUC = \sum_{i=0}^{x} \left( \frac{NPRS_i + NPRS_{i+1}}{2} \right) * (T_{i+1} - T_i)$$

Where: NRS<sub>i</sub> = NRS at rest at time I, and  $(T_{i+1} - T_i)$  is the Time difference in hours between time i and time i+1.

Missing NRS will be handled as discussed in Section 7.1. AUC values will be analyzed using a 1-factor (treatment) analysis of variance (ANOVA) model with treatment as the main effect.

The AUC analyses will be presented in a summary table with standard summary statistics for each treatment group as well as active vs. placebo mean differences, standard errors, confidence intervals and comparison p-values as appropriate. In addition, AUC<sub>0-96h</sub> at rest will be analyzed using Wilcoxon sum-rank test.


Statistical Analysis Plan Protocol Number: CA-PS-203 Date: 24APR2019

The individual NRS and the computed AUC variables will be listed for all individual subjects.

# 7.4.4 Opioid Free (OF) 0-96h (Secondary Efficacy Endpoint)

Opioid use is recorded on the rescue medication eCRF from the end of surgery through the D15 follow up/Early termination (ET). If additional opioids, other than the study rescue medications, appear on the concomitant medications page and can be identified, those opioids will also be considered.

The percentage of subjects who do not require opioids (are Opioid Free or OF) will be analyzed using a logistic regression with treatment group as the main effect. The analysis will compare the odds ratios of the proportions of OF subjects between each treatment group and the placebo group. A summary of frequencies as well as odds ratio, 95% confidence intervals and p-values will be presented for 0 to 96 hours (OF<sub>0 to 96h</sub>).

#### 7.4.5 Total Opioid Consumption (OC) in Daily Oral Morphine equivalents 0-96h (Secondary Efficacy Endpoint)

The amount of opioids taken as rescue will be calculated using the rescue medication page of the eCRF. If additional opioids, other than the study rescue medications, appear on the concomitant medications page and can be identified, those opioids will also be included (in terms of morphine equivalents) in the total consumed. Table 3 will be used to calculate the morphine equivalent dose (MED) for each medication. The total opioid consumption for each day for each subject will be calculated as the sum of the MEDs of all of the medications taken on that day. For example, if a subject takes 5 MED morphine on Day 1 and Day 2, and 10 MED of Oxycodone on Day 2, the total consumption for Day 1 is 5 MED, and the total consumption for Day 2 is 15 MED. Subjects that take no opioids on a day will have a total opioid consumption value of zero for that day.


Table 3 Equianalgesic Conversion Table

| Opioid (Doses in mg) | Conversion Factor to IV morphine | Conversion Factor to PO morphine |
|---|---|---|
| IV Fentanyl | 100 | |
| IV Hydromorphone | 6 | |
| IV Morphine | 1 | 6* |
| PO Hydrocodone | | 1 |
| PO Morphine | | 1 |
| PO Oxycodone | | 1.5 |
| PO Tramadol | | 0.1 |

For any IV opioid, we will use a 2-step process to calculate its oral (PO) morphine equivalent dose (MED):

- 1. Convert its IV dose to IV morphine MED by multiplying by the conversion factor for IV equivalence.
- 2. Once the IV morphine MED is calculated, convert to the PO morphine MED using the conversion factor for PO equivalence.

For any PO opioid, use the conversion factor to calculate the PO MED.

\*Note that for non-tolerant patients, we are using the 6:1 conversion for IV to PO morphine.

Total opioid consumption will be calculated for 0-96 hours ( $OC_{0 \text{ to 96h}}$ ). An ANOVA with treatment arm as the main effect will be performed. A separate summary containing only subjects that have taken at least one dose of rescue will be performed if warranted.

#### 8. SAFETY EVALUATION

#### 8.1 Overview of Safety Analysis Methods

All safety outcomes will be summarized using the safety population. No formal statistical comparisons will be performed for safety outcomes. Safety outcomes include:

- Incidence of spontaneous reported treatment-emergent adverse events (TEAEs) or serious adverse events (SAEs)
- Physical examination (PE)


- Vital signs
- Surgical site assessments
- Neurosensory testing near the incision
- X-ray of the operated knee
- Rebound or worsening pain
- ECG
- Clinical laboratory test results

#### 8.2 Adverse Events and SAEs

All AEs and SAEs are documented and followed from the time the subject have signed the informed consent form (ICF) until Day 29 or later as necessary. AEs will be coded by system organ class (SOC) and preferred term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA Version 21.0) reporting system. All coding will be reviewed prior to database lock. All recorded AEs will be listed, but only TEAEs will be summarized.

Treatment-emergent AEs are defined as any of the following:

- Non-serious AEs with onset on the date of treatment with the study drug through Day 29
  or Early Termination, whichever occurs first.
- Serious AEs with onset on the date of treatment with the study drug through 30 days after Day 29 or Early Termination, whichever occurs first.
- AEs that start before the start of treatment but increase in severity or relationship at the time of or following the start of treatment through Day 29 or Early Termination, whichever occurs first.

For evaluation of causal relatedness to treatment, the categories are probably related, possibly related or unlikely related. For categorization in the summary tables, AEs designated as probably or possibly related will be considered to be related.

For the evaluation of event severity terms, the criteria are mild, moderate, severe or potentially life-threatening. In addition to a listing of all TEAEs, treatment related TEAEs, serious TEAEs, Deaths, and TEAEs leading to premature discontinuation from the study will be provided.


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

An overall summary will be prepared giving for each treatment group and overall both the number of TEAEs, and the number of subjects with at least one TEAEs, as well as SAEs, treatment related TEAEs and TEAEs leading to premature discontinuation from study.

The number of subjects with AEs will be summarized for each treatment group by SOC and PT sorted in alphabetically by SOC, and then by PT within SOC. These summaries will be given by treatment in separate tables for each of the following TEAE event sets:

- All events
- Treatment related events
- Serious events
- Events leading to premature discontinuation from study
- Events by maximum severity

If a given subject experiences a TEAE that maps to the same PT/SOC more than once, the subject will be counted only once for the SOC/PT at the greatest severity (i.e., mild, moderate, or severe) and causality (i.e., attribution to study material).

Duration of a TEAE lasting more than 24 hours will be computed in days as the stop date of the event minus the start date plus 1 and will be reported in days. TEAEs lasting less than 24 hours will be computed as stop date/time minus start date/time. If reported as ongoing at the time of database lock, the stop date is defined as the date of the last visit or the last date of any event for the subject in the database, whichever is later.

If a TEAE is considered resolved, but the stop date is missing, the last day of the month will be imputed if the month and year are available. If only the year is available, and the year is the same as the year of the last visit, the stop date will be the latest of the last visit date or latest event for the subject in the database.

If the year of the event is prior to the year of the last treatment, the end day and month will be set to 31 December.

For missing or partial start and stop dates/times, the most conservative imputation will be used (AEs will be assumed to be temporally related to the study medication). <u>Table 4</u> will be used to impute any missing dates/times:


Table 4 Table of Imputation Rules for Missing AE Start Dates

| Missing Date<br>Portion | Prior to<br>Treatment | Same as Treatment<br>Start Date | After Treatment Start<br>Date |
|---|---|---|---|
| Day | Month and Year <<br>Month and Year of<br>Study treatment: | Month and Year =<br>Month and Year of<br>Study treatment: | Month and Year ><br>Month and Year of<br>Study Treatment: |
| | Start Day = 1 Stop Day=last day of | Start Day = Day of first<br>treatment | Start Day = 1<br>Stop Day=last day of |
| the month | | Stop Day= last day of the month | the month |
| Day and Month<br>Define Day as | Year < Year of first treatment: | Year = Year of study<br>treatment: | Year > Year of study treatment: |
| above, then: | Start Month = July | Start Month = Month of<br>study treatment | Start Month = January |
| | Stop Month = Dec | Stop Month = Dec | Stop Month = Dec |
| Day, Month, and<br>Year | · · | | |
| Time | Missing start times will be imputed as 00:01 | | |
| | Missing stop times will be imputed as 23:59 | | |

After following these imputation rules, if the start date/time is imputed as a date after the end date/time, the start date/time will be set to the end date/time to provide a positive duration for the event incidence.

Missing assessments for AE study medication relationship or severity will be analyzed as related or severe respectively. No other imputation is planned for safety data.

## 8.3 Physical Examination

A complete medical history and physical examination including all major body systems will be performed at Screening. In addition, a focused interim medical history and targeted physical examination will be performed prior to surgery (if not done on D-1), and to capture changes after Surgery, at 96 hours (± 4 hours) after the administration of study medication, but prior to discharge, and Days 8, 15 and 29/ET after the administration of study medication.

CONFIDENTIAL


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

Abnormal or clinically significant physical exam will be recorded as AEs. Physical examination results will be listed for individual subjects.

## 8.4 Vital Signs

Vital signs results including blood pressure (systolic and diastolic; mmHg), heart rate (beats per minute), respiration rate (breaths/min), and temperature will be listed for individual subjects.

Baseline for vital signs measurements will be defined as the last evaluation before dosing with study medication. Summary statistics, including change from baseline, will be determined for each measure and will be summarized by treatment and time point.

## 8.5 Surgical Site Assessments and Rebound (or Worsening) Pain Assessments

Surgical sites will be assessed at 96 hours (prior to discharge from the unit) and then as an outpatient on Days 8, 15 and 29. The investigator will evaluate their satisfaction with the healing of the wound during this surgical site assessment using an 11-point scale (0- 10) where a score of 0 is "completely unsatisfied" and a score of 10 is "completely satisfied). In addition, subjects will report whether they have noted any worsening pain (rebound pain; Y/N) at the surgical site since the prior visit at Days 8, 15 and/or 29.

All data will be presented in data listings. Results of surgical site assessments and the number of subjects with rebound pain will be summarized descriptively by treatment and time point.

#### 8.6 Neurosensory Test

Neurosensory testing near the incision (compared to a similar site on the opposite leg) will be performed at screening, T96h (prior to discharge from the unit) and then as an outpatient on Days 8, 15, and 29.

The neurosensory assessment results will be listed and the number of subjects in each response will be summarized descriptively by treatment and time point by wound (cephalad or caudad).

# 8.7 X-ray of the Operated Knee

X-ray of the operated knee on Day 29 and later if any evidence of abnormal bone healing until resolution or stabilization. Also perform this at early termination if subject gives consent.


Protocol Number: CA-PS-203 Date: 24APR2019

Statistical Analysis Plan

Results of x-ray of the operated knee will not be entered in database. Date and time of x-ray performed will be listed.

#### 8.8 ECG

ECG examination will be assessed at screening and 24 hours (±2 hours) after study medication administration.

12-Lead ECGs will be performed after the subject has been resting in a recumbent/supine position for at least 5 minutes. ECGs will be signed and dated by a medically-qualified individual to confirm review of the ECG and verify whether any abnormalities are clinically significant.

Number of subjects with abnormal results will also be summarized by treatment and time point.

# 8.9 Clinical Laboratory Test Results

Clinical laboratory tests (chemistry, hematology/coagulation and urinalysis) will be collected at screening and before discharge from the inpatient unit (T96h). All results will be listed. For each lab test, the raw value and change from screening will be summarized by treatment.

Each clinical laboratory test will be defined by the clinical laboratory to be "Low", "Normal", or "High", according to the normal reference range from the clinical laboratory.

The number and percentage of subjects who have a shift from within to outside the normal reference range from screening to T96h will be summarized by treatment.

#### 8.10 Drugs of Abuse and Alcohol Screens, Pregnancy Test

Pregnancy (for female subjects of childbearing potential), urine drug screen and alcohol (breath or saliva) tests will be performed at screening and pre-surgery.

Results will be listed for individual subjects. Each test result will be defined to be "negative" or "positive".

#### 8.11 Subject pain Assessment Training and Surgery Details

Pain assessment training will be provided during screening. Subjects will re-watch video prior to surgery. Patient pain assessment training and surgery Details will be documented in CRFs and will be listed for each subject.


Statistical Analysis Plan Protocol Number: CA-PS-203 Date: 24APR2019

## 9. PHARMACOKINETIC EVALUATION

The time points for PK whole blood collections will be at baseline (from Check-in and up to 30 min prior to surgery), 5, 10, 15, 30, 45 minutes, and at hours 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 30, 36 and 48 (for a total of 20 samples) after the end of study treatment administration.

Actual sampling times will be used to calculate plasma-derived PK parameters. Full details of PK endpoints/analyses will be described in a separate PK Analysis plan.

#### 10. OTHER ANALYSES

All additional analyses of Pilot Stage data not included in this SAP, conducted after Pilot stage unblinding will be considered exploratory and will be presented and identified separately in the CSR.

#### 11. INTERIM ANALYSES

An interim unblinded analysis may be performed after the last subject from each pilot stage cohort has completed the D8 visit. Since no Stage 2 data will be collected, final data from the initial Pilot stage will be summarized and no additional SAP or analyses will be performed...

#### 12. REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583.

US Federal Register. (1996) International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320.

Guidance for Industry (2014) Analgesic Indications: Developing Drug and Biological Products -Draft Guidance. Department of Health and Human Services: Food and Drug Administration. Center for Drug Evaluation and Research (CDER) February 2014 Clinical/Medical.


# 13. APPENDICES

# 13.1 Planned Tables, Figures and Listings

# 13.1.1 Tables

| | T | |
|---|---|---|
| Table 14.1.1 | All Subjects | Summary of Subject Disposition |
| Table 14.1.2 | Randomized | Summary of Protocol Deviations |
| | Subjects | |
| Table 14.1.3 | Safety | Summary of Demographics and Baseline Characteristics |
| | Population | |
| Table 14.1.4 | Safety | Summary of Concomitant Medications by ATC Class and |
| | Population | Preferred Term |
| Table 14.1.5 | Safety | Summary of Subject NRS and NRS at Rescue Diary Compliance |
| | Population | |
| Table 14.2.1 | Safety | ANOVA Analysis of Hour 96 NRS at Rest – WOCF (Primary Analysis) |
| | Population | |
| Table 14.2.1.1 | Safety | Wilcoxon Analysis of Hour 96 NRS at Rest – WOCF |
| | Population | · |
| Table 14.2.2.1 | Safety | ANOVA Analysis of NRS at Rest by Hour |
| | Population | |
| Table 14.2.2.2 | Safety | ANOVA Analysis of NRS at Rest by Morning/Night |
| | Population | |
| Table 14.2.2.3 | Safety | Wilcoxon Analysis of NRS at Rest by Hour |
| T 11 44004 | Population | MULL A L.: CNDO (D. (L. M: WILL) |
| Table 14.2.2.4 | Safety | Wilcoxon Analysis of NRS at Rest by Morning/Night |
| Table 14.2.3 | Population | ANOVA Analysis of AUC (0-96) NRS at Rest – WOCF (Secondary |
| 1 4.2.3 | Safety<br>Population | Efficacy Analysis) |
| Table 14.2.3.1 | Safety | Wilcoxon Analysis of AUC (0-96) NRS at Rest - WOCF |
| 1 4.2.3.1 | Population | Wilcoxoff Affaiysis of AOC (0-90) NNS at Nest - WOCI |
| Table 14.2.4 | Safety | Logistic Analysis of Proportion of Subjects Who Are Opioid Free |
| 1 4 4 1 1 1 1 | Population | (Secondary Efficacy Analysis) |
| Table 14.2.5 | Safety | ANOVA Analysis of Opioid Consumption (in Morphine Equivalents) |
| 1 4510 1 112.0 | Population | (Secondary Efficacy Analysis) |
| Table 14.3.1 | Safety | Overall Summary of Treatment-Emergent Adverse Events (TEAEs) |
| 1 3010 1 110.1 | Population | Total Gallinary of Froduition Emorgon Advoice Evente (FEAEs) |
| Table 14.3.1.1 | Safety | Summary of Treatment-Emergent Adverse Events (TEAEs) by System |
| 1 4010 14.0.1.1 | Population | organ Class and Preferred Term |
| Table 14.3.1.2 | Safety | Summary of Treatment Related Treatment-Emergent Adverse Events |
| 14510 17.0.1.2 | Population | (TEAEs) by System organ Class and Preferred Term |
| Table 14.3.1.3 | Safety | Summary of Serious Adverse Events by System organ Class and |
| 1 4016 14.0.1.0 | Population | Preferred Term |
| Table 14.3.1.4 | • | Summary of Treatment-Emergent Adverse Events (TEAEs) Leading to |
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | Safety | Study Discontinuation by System organ Class and Preferred Term |
| Table 14.3.1.5 | Population | Summary of Treatment-Emergent Adverse Events (TEAEs) by System |
| 1 4.3.1.5 | Safety | organ Class, Preferred Term and Severity |
| | Population | organ Olass, Freiened Ferni and Oevenly |


| Table 14.3.1.6Safety PopulationSummary of Treatment-Emergent Adverse Events (TEAEs) by System organ Class, Preferred Term and Relationship to Study DrugTable 14.3.2.1Safety PopulationSummary of Chemistry Laboratory Tests: Results and Change from BaselineTable 14.3.2.2Safety PopulationSummary of Chemistry Laboratory Tests: Shift from BaselineTable 14.3.3.1Safety PopulationSummary of Coagulation Laboratory Tests: Results and Change from BaselineTable 14.3.4.1Safety PopulationSummary of Coagulation Laboratory Tests: Shift from BaselineTable 14.3.4.2Safety PopulationSummary of Hematology Laboratory Tests: Results and Change from BaselineTable 14.3.5.1Safety PopulationSummary of Hematology Laboratory Tests: Shift from BaselineTable 14.3.5.2Safety PopulationSummary of Urinalysis Laboratory Tests: Results and Change from BaselineTable 14.3.6Safety PopulationSummary of Urinalysis Laboratory Tests: Shift from BaselineTable 14.3.7Safety PopulationSummary of Vital Signs: Results and Change from BaselineTable 14.3.8Safety PopulationSummary of Surgical Site AssessmentTable 14.3.9.1Safety PopulationSummary of Neurosensory Exam – Cephalad to WoundTable 14.3.9.2Safety PopulationSummary of Neurosensory Exam – Caudad to WoundTable 14.3.10Safety PopulationSummary of ECG Exam Abnormal Findings | | , | |
|---|---|---|---|
| Table 14.3.2.1 Safety Population Table 14.3.2.2 Safety Population Table 14.3.3.1 Safety Population Table 14.3.3.1 Safety Population Table 14.3.3.2 Safety Population Table 14.3.3.2 Safety Population Table 14.3.3.2 Safety Population Table 14.3.3.2 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.5.2 Safety Population Table 14.3.5.2 Safety Population Table 14.3.5.3 Safety Population Table 14.3.5 Safety Population Table 14.3.5 Safety Population Table 14.3.5 Safety Population Table 14.3.5 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9 Safety Population Table 14.3.9 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound | Table 14.3.1.6 | Safety | Summary of Treatment-Emergent Adverse Events (TEAEs) by System |
| Population Baseline | | Population | organ Class, Preferred Term and Relationship to Study Drug |
| Table 14.3.2.2 Safety Population Table 14.3.3.1 Safety Population Table 14.3.3.2 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.3 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.3 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.3 Safety Population Table 14.3.9.3 Safety Population Table 14.3.9.1 Safety Population | Table 14.3.2.1 | Safety | Summary of Chemistry Laboratory Tests: Results and Change from |
| Population Table 14.3.3.1 Safety Population Safety Populat | | Population | Baseline |
| Table 14.3.3.1 Safety Population Table 14.3.3.2 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.3 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.10 Safety Population Table 14.3.10 Safety Population Table 14.3.10 Safety | Table 14.3.2.2 | Safety | Summary of Chemistry Laboratory Tests: Shift from Baseline |
| Table 14.3.3.2 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9 Safety Population Table 14.3.9 Safety Population Table 14.3.8 Safety Population Table 14.3.9 Safety Summary of Neurosensory Exam – Cephalad to Wound Population Table 14.3.9 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.9 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.3.2 Safety Population Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9 Safety Summary of Neurosensory Exam – Cephalad to Wound Table 14.3.9 Safety Population Table 14.3.9 Safety Summary of Neurosensory Exam – Caudad to Wound Table 14.3.9 Safety Summary of Neurosensory Exam – Caudad to Wound Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | Table 14.3.3.1 | Safety | Summary of Coagulation Laboratory Tests: Results and Change from |
| Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound | | Population | Baseline |
| Table 14.3.4.1 Safety Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Population Summary of Hematology Laboratory Tests: Shift from Baseline Summary of Urinalysis Laboratory Tests: Shift from Baseline Summary of Vital Signs: Results and Change from Baseline Summary of Vital Signs: Results and Change from Baseline Summary of Surgical Site Assessment Summary of Rebound Pain Assessment Summary of Neurosensory Exam – Cephalad to Wound Summary of Neurosensory Exam – Caudad to Wound Summary of Neurosensory Exam – Caudad to Wound Summary of ECG Exam Abnormal Findings | Table 14.3.3.2 | Safety | Summary of Coagulation Laboratory Tests: Shift from Baseline |
| Population Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety | | Population | |
| Table 14.3.4.2 Safety Population Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.8 Safety Population Table 14.3.9 Safety Population Table 14.3.8 Safety Population Table 14.3.9 Safety Summary of Neurosensory Exam – Cephalad to Wound Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Caudad to Wound Table 14.3.10 Safety Summary of Surgical Site Assessment Summary of Neurosensory Exam – Caudad to Wound | Table 14.3.4.1 | Safety | Summary of Hematology Laboratory Tests: Results and Change from |
| Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Summary of Neurosensory Exam – Caudad to Wound Population Summary of Neurosensory Exam – Caudad to Wound Population Summary of Neurosensory Exam – Caudad to Wound Population Summary of Neurosensory Exam – Caudad to Wound Population Summary of Summary of Neurosensory Exam – Caudad to Wound Population Summary of Summary of Summary of Neurosensory Exam – Caudad to Wound Population Summary of ECG Exam Abnormal Findings | | Population | Baseline |
| Table 14.3.5.1 Safety Population Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.3 Safety Population Table 14.3.9.4 Safety Population Table 14.3.9.5 Safety Population Table 14.3.9.7 Safety Population Table 14.3.9.8 Safety Population Table 14.3.9.9 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | Table 14.3.4.2 | Safety | Summary of Hematology Laboratory Tests: Shift from Baseline |
| Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of Summary of Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.5.2 Safety Population Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Population Summary of Vital Signs: Results and Change from Baseline Summary of Surgical Site Assessment Population Summary of Rebound Pain Assessment Summary of Rebound Pain Assessment Population Summary of Neurosensory Exam – Cephalad to Wound Population Summary of Neurosensory Exam – Caudad to Wound Population Summary of Summary of Summary of Neurosensory Exam – Caudad to Wound Population Summary of Summary | Table 14.3.5.1 | Safety | |
| Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Cephalad to Wound Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | Baseline |
| Table 14.3.6 Safety Population Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Cephalad to Wound Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | Table 14.3.5.2 | Safety | Summary of Urinalysis Laboratory Tests: Shift from Baseline |
| Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Cephalad to Wound Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.7 Safety Population Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Summary of ECG Exam Abnormal Findings | Table 14.3.6 | Safety | Summary of Vital Signs: Results and Change from Baseline |
| Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Cephalad to Wound Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.8 Safety Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | Table 14.3.7 | Safety | Summary of Surgical Site Assessment |
| Population Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.9.1 Safety Population Table 14.3.9.2 Safety Population Table 14.3.10 Safety Summary of Neurosensory Exam – Caudad to Wound Population Summary of Neurosensory Exam – Caudad to Wound Population Summary of ECG Exam Abnormal Findings | Table 14.3.8 | Safety | Summary of Rebound Pain Assessment |
| Population Table 14.3.9.2 Safety Summary of Neurosensory Exam – Caudad to Wound Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.9.2 Safety Population Summary of Neurosensory Exam – Caudad to Wound Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | Table 14.3.9.1 | Safety | Summary of Neurosensory Exam – Cephalad to Wound |
| Population Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | | Population | |
| Table 14.3.10 Safety Summary of ECG Exam Abnormal Findings | Table 14.3.9.2 | Safety | Summary of Neurosensory Exam – Caudad to Wound |
| | | Population | |
| Population | Table 14.3.10 | Safety | Summary of ECG Exam Abnormal Findings |
| | | Population | |


# 13.1.2 Listings

| Listing 16.2.2 All Subjects Eligibility Listing 16.2.5 All Subjects Protocol Deviations Listing 16.2.6 All Subjects Subject Subject disposition/ Early Termination Listing 16.2.6 All Randomized Subjects Demographics and Baseline Characteristics Listing 16.2.7 All Randomized Subjects Prior and Concomitant Medications Listing 16.2.8.1 All Randomized Subjects Prior and Concomitant Medications Listing 16.2.8.2 All Randomized Subjects Rescue Medication Therapies Listing 16.2.8.3 All Randomized Subjects Surgery Listing 16.2.10 All Randomized Subjects Subjects Surgery Listing 16.2.11 All Randomized Subjects Subject | | | , |
|---|---|---|---|
| Listing 16.2.4 All Subjects Protocol Deviations Listing 16.2.5 All Subjects Subject disposition/ Early Termination Listing 16.2.6 All Randomized Subjects Demographics and Baseline Characteristics Listing 16.2.7 All Randomized Subjects Prior and Concomitant Medications Listing 16.2.8.1 All Randomized Subjects Prior and Concomitant Medications Listing 16.2.8.2 All Randomized Subjects Rescue Medication Administration Listing 16.2.9 All Randomized Subjects Surgery Listing 16.2.10 All Randomized Subjects Surgery Listing 16.2.11 All Randomized Subjects Subject Sutdy Drug Administration, Pain Assessment Training and Discharge Listing 16.2.12.1 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Pisiting 16.2.12.2 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.13 All Randomized Subjects Pain Intensity Assessment (NRS with Ambulation) Listing 16.2.14 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.16.1 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.16.1 All Randomized Subjects (NOOS - ADL Listing 16.2.16.2 All Randomized Subjects (NOOS - ADL Listing 16.2.16.3 All Randomized Subjects (NOOS - Pain Listing 16.2.16.4 All Randomized Subjects (NOOS - Pain Listing 16.2.17.1 All Randomized Subjects (NOOS - Pain Listing 16.2.17.2 All Randomized Subjects (NOOS - Pain Listing 16.2.17.3 All Randomized Subjects (NOOS - Quality of Life Listing 16.2.17.3 All Randomized Subjects (NOOS - Quality of Life Listing 16.2.17.3 All Randomized Subjects (NOOS - Quality of Life Listing 16.2.18.3 All Randomized Subjects (NOOS - Port Rec Listing 16.2.18.4 All Randomized Subjects (NOOS - Quality of Life Listing 16.2.18.4 All Randomized Subjects (NOOS - Quality of Life Listing 16.2.18.4 All Randomized Subjects (NOOS - Port Results Listing 16.2.18.4 All Randomized Subjects (NOOS - Port Results Listing 16.2.20 All Randomized Subjects (NOOS - Port Results Listing 16.2.21 All Randomized Subjects (NOOS - Port Results Listing 16.2.22 All Randomized Subjects (NOOS - | Listing 16.2.1 | All Subjects | Randomization and Study Population |
| Listing 16.2.4 All Subjects Subject (Isting 16.2.5 All Randomized Subjects Listing 16.2.6 All Randomized Subjects Disting 16.2.8.1 All Randomized Subjects (Isting 16.2.8.1 All Randomized Subjects Prior and Concomitant Medications Listing 16.2.8.2 All Randomized Subjects Rescue Medication Administration Non-Medication Therapies All Randomized Subjects Surgery All Randomized Subjects Surgery (Isting 16.2.9 All Randomized Subjects Surgery Subjects All Randomized Subjects Surgery (Isting 16.2.10 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.1.1 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Subjects (Isting 16.2.1.2 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Pain Intensity Assessment (NRS at Rest) Pain Intensity Assessment (NRS with Ambulation) (Isting 16.2.1.3 All Randomized Subjects List of Efficacy Endpoints (Isting 16.2.1.6 All Randomized Subjects (Investigator Global Evaluation (PGE) (Investigator Global Evaluation (IGE) (Investigator Global Evaluation (IGE) (Isting 16.2.16.2 All Randomized Subjects (Investigator Global Evaluation (IGE) (Isting 16.2.16.3 All Randomized Subjects (Investigator Global Evaluation (IGE) (Isting 16.2.16.3 All Randomized Subjects (Investigator Global Evaluation (IGE) (Isting 16.2.16.4 All Randomized Subjects (Isting 16.2.16.5 All Randomized Subjects (Isting 16.2.16.5 All Randomized Subjects (Isting 16.2.17.1 All Randomized Subjects (Isting 16.2.17.2 All Randomized Subjects (Isting 16.2.17.3 All Randomized Subjects (Isting 16.2.17.4 All Randomized Subjects (Isting 16.2.18.1 All Randomized Subjects (Isting 16.2.18.3 All Randomized Subjects (Isting 16.2.18.3 All Randomized Subjects (Isting 16.2.18.3 All Randomized Subjects (Isting 16.2.18.3 All Randomized Subjects (Isting 16.2.18.4 All Randomized Subjects (Isting 16.2.18.4 All Randomized Subjects (Isting 16.2.20 All Randomized Subjects (Isting 16.2.20 All Randomized Subjects (Isting 16.2.20 All Randomized Subjects (Isting 16.2.20 All Randomized Subjects ( | Listing 16.2.2 | All Subjects | Informed Consent and Re-Consent |
| Listing 16.2.5 All Subjects Subject disposition/ Early Termination Listing 16.2.6 All Randomized Subjects Demographics and Baseline Characteristics Listing 16.2.7 All Randomized Subjects Medical/ Surgical History Listing 16.2.8.1 All Randomized Subjects Prior and Concomitant Medications Listing 16.2.8.2 All Randomized Subjects Rescue Medication Administration Listing 16.2.8.3 All Randomized Subjects Rescue Medication Administration Listing 16.2.9 All Randomized Subjects Surgery Listing 16.2.10 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.1.1 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.1.2.1 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.1.2.1 All Randomized Subjects Pain Intensity Assessment (NRS with Ambulation) Listing 16.2.1.3 All Randomized Subjects List of Efficacy Endpoints Listing 16.2.1.4 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.1.5 All Randomized Subjects Investigator Global Evaluation (IGE) Listing 16.2.1.6.1 All Randomized Subjects KOOS - Knee Symptoms Listing 16.2.1.6.2 All Randomized Subjects KOOS - ADL Listing 16.2.1.6.3 All Randomized Subjects KOOS - Pain Listing 16.2.1.6.4 All Randomized Subjects KOOS - Sport/ Rec Listing 16.2.1.6.5 All Randomized Subjects KOOS - Quality of Life Listing 16.2.1.6.5 All Randomized Subjects Adverse Events Listing 16.2.1.7.1 All Randomized Subjects Serious Adverse Events Listing 16.2.1.7.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.1.7.3 All Randomized Subjects Serious Adverse Events Listing 16.2.1.7.4 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.1.8.3 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.1.8.4 All Randomized Subjects Demonstry Laboratory Test Results Listing 16.2.1.8.4 All Randomized Subjects Demonstry Laboratory Test Results Listing 16.2.2.1 All Randomized Subjects Demonstry Laboratory Test Results Listing 16.2.2.1 All Randomized Subject | Listing 16.2.3 | All Subjects | |
| Listing 16.2.6 Listing 16.2.7 All Randomized Subjects Medical/ Surgical History Listing 16.2.8.1 All Randomized Subjects Medical/ Surgical History Prior and Concomitant Medications Listing 16.2.8.2 All Randomized Subjects Rescue Medication Administration Non-Medication Therapies Listing 16.2.9 All Randomized Subjects Surgery Listing 16.2.10 All Randomized Subjects Surgery Listing 16.2.11 All Randomized Subjects Surgery Listing 16.2.1.1 All Randomized Subjects Subjects NRS and NRS at Rescue Diary Compliance Listing 16.2.1.2 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.1.2 All Randomized Subjects Pain Intensity Assessment (NRS with Ambulation) Listing 16.2.1.3 All Randomized Subjects List of Efficacy Endpoints Listing 16.2.1.4 All Randomized Subjects Listing 16.2.1.5 All Randomized Subjects Listing 16.2.1.6 Listing 16.2.1.6 All Randomized Subjects Listing 16.2.1.6 Listing 16.2.1.6 All Randomized Subjects Listing 16.2.1.6 All Randomized Subjects KOOS - Knee Symptoms Listing 16.2.1.6 All Randomized Subjects KOOS - Pain Listing 16.2.1.6 All Randomized Subjects KOOS - Pain Listing 16.2.1.7 All Randomized Subjects KOOS - Pain Listing 16.2.1.7 All Randomized Subjects KOOS - Pain Listing 16.2.1.7 All Randomized Subjects KOOS - Quality of Life Listing 16.2.1.7 All Randomized Subjects COS - Quality of Life Listing 16.2.1.7 All Randomized Subjects Listing 16.2.1.7 All Randomized Subjects Consultity of Life Listing 16.2.1.7 All Randomized Subjects Listing 16.2.1.7 All Randomized Subjects Computed Adverse Events Listing 16.2.1.8 All Randomized Subjects Listing 16.2.1.8 All Randomized Subjects Consultity of Life Adverse Events Listing 16.2.1.8 All Randomized Subjects Consultity of Life Adverse Events Listing 16.2.1.8 All Randomized Subjects Consultity of Life Adverse Events Listing 16.2.1.8 All Randomized Subjects Consultity of Life Adverse Events Listing 16.2.1.8 All Randomized Subjects Consultity of Life Adverse Events Listing 16.2.1.8 All Randomized Subjects Consultity of Life Adverse | Listing 16.2.4 | | |
| Listing 16.2.8.1 All Randomized Subjects Listing 16.2.8.2 All Randomized Subjects Listing 16.2.8.3 All Randomized Subjects Listing 16.2.8.3 All Randomized Subjects Listing 16.2.9 All Randomized Subjects Listing 16.2.10 All Randomized Subjects Listing 16.2.11 All Randomized Subjects Listing 16.2.11 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.2 All Randomized Subjects Listing 16.2.12.3 All Randomized Subjects Listing 16.2.13 All Randomized Subjects Listing 16.2.14 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.4 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.4 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.17.1 All Randomized Subjects Listing 16.2.17.2 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.5 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.19.4 All Randomized Subjects Listing 16.2.19.4 All Randomized Subjects Listing 16.2.19.4 All Randomized Subjects Listing 16.2.19.4 All Randomized Subjects Listing 16.2.19.4 All Randomized Subjects Listing 16.2.20 All Randomized Subjects Listing 16.2.21 All Randomized Subjects Listing 16.2.22 All Randomized Subjects Listing 16.2.23 All Randomized Subjects Listing 16.2.24 All Randomized Subjects Listing 16.2.25 A | Listing 16.2.5 | All Subjects | Subject disposition/ Early Termination |
| Listing 16.2.8.1 All Randomized Subjects Rescue Medication Administration Listing 16.2.8.3 All Randomized Subjects Rescue Medication Administration Listing 16.2.9 All Randomized Subjects Non-Medication Therapies Listing 16.2.10 All Randomized Subjects Surgery Listing 16.2.11 All Randomized Subjects Subjects Non-Medication Therapies Listing 16.2.12 All Randomized Subjects Subjects NRS and NRS at Rescue Diary Compliance Listing 16.2.1.1 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.1.2 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.1.3 All Randomized Subjects Pain Intensity Assessment (NRS with Ambulation) Listing 16.2.1.4 All Randomized Subjects Investigator Global Evaluation (PGE) Listing 16.2.1.5 All Randomized Subjects Investigator Global Evaluation (IGE) Listing 16.2.1.6.1 All Randomized Subjects KOOS - Rnee Symptoms Listing 16.2.1.6.2 All Randomized Subjects KOOS - Pain Listing 16.2.1.6.3 All Randomized Subjects KOOS - Pain Listing 16.2.1.6.4 All Randomized Subjects KOOS - Pain Listing 16.2.1.6.5 All Randomized Subjects KOOS - Quality of Life Listing 16.2.1.7.1 All Randomized Subjects KOOS - Quality of Life Listing 16.2.1.7.2 All Randomized Subjects Serious Adverse Events Listing 16.2.1.7.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.1.7.3 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.1.8.1 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.1.8.2 All Randomized Subjects Demistry Laboratory Test Results Listing 16.2.2.1 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.2.1 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.1 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.1 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.2 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Results Listing 16.2 | Listing 16.2.6 | All Randomized Subjects | Demographics and Baseline Characteristics |
| Listing 16.2.8.2 All Randomized Subjects Listing 16.2.8.3 All Randomized Subjects Listing 16.2.9 All Randomized Subjects Surgery Listing 16.2.10 All Randomized Subjects Listing 16.2.11 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.13 All Randomized Subjects Listing 16.2.14 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.16 All Randomized Subjects Listing 16.2.16 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.4 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.17.1 All Randomized Subjects Listing 16.2.17.2 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.5 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.18.2 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.5 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.18.2 All Randomized Subjects Listing 16.2.18.2 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.5 All Randomized Subjects Listing 16.2.2.8 All Randomized Subjects Listing 16.2.2.9 All Randomized Subjects Listing 16.2.2.1 All Randomized Subjects Listing 16.2.2.2 All Randomized Subjects Listing 16.2.2.3 All Randomized Subjects Listing 16.2.2.4 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing | Listing 16.2.7 | All Randomized Subjects | Medical/ Surgical History |
| Listing 16.2.8.3 All Randomized Subjects Listing 16.2.9 All Randomized Subjects Surgery Listing 16.2.11 All Randomized Subjects Listing 16.2.12 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.2 All Randomized Subjects Listing 16.2.12.2 All Randomized Subjects Listing 16.2.13 All Randomized Subjects Listing 16.2.14 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.4 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.17.1 All Randomized Subjects Listing 16.2.17.2 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.18.2 All Randomized Subjects Listing 16.2.18.3 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.2.19 All Randomized Subjects Listing 16.2.2.2 All Randomized Subjects Listing 16.2.2.3 All Randomized Subjects Listing 16.2.2.4 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 1 | Listing 16.2.8.1 | All Randomized Subjects | Prior and Concomitant Medications |
| Listing 16.2.9 All Randomized Subjects Listing 16.2.10 All Randomized Subjects Listing 16.2.11 All Randomized Subjects Listing 16.2.12.1 All Randomized Subjects Listing 16.2.12.2 All Randomized Subjects Listing 16.2.12.2 All Randomized Subjects Listing 16.2.13 All Randomized Subjects Listing 16.2.14 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.4 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.17.1 All Randomized Subjects Listing 16.2.17.2 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.5 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.5 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.2.1 All Randomized Subjects Listing 16.2.2.1 All Randomized Subjects Listing 16.2.2.1 All Randomized Subjects Listing 16.2.2.2 All Randomized Subjects Listing 16.2.2.3 All Randomized Subjects Listing 16.2.2.4 All Randomized Subjects Listing 16.2.2.5 All Randomized Subjects Listing 16.2. | Listing 16.2.8.2 | All Randomized Subjects | Rescue Medication Administration |
| Listing 16.2.10 All Randomized Subjects Listing 16.2.11 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.12.1 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.13 All Randomized Subjects Pain Intensity Assessment (NRS with Ambulation) Listing 16.2.14 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Investigator Global Evaluation (IGE) Listing 16.2.16.2 All Randomized Subjects KOOS - Knee Symptoms Listing 16.2.16.3 All Randomized Subjects KOOS - ADL Listing 16.2.16.4 All Randomized Subjects KOOS - Pain Listing 16.2.16.5 All Randomized Subjects KOOS - Pain Listing 16.2.16.5 All Randomized Subjects KOOS - Pain Listing 16.2.17.1 All Randomized Subjects KOOS - Pain Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Serious Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Listing 16.2.18.1 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.2.1 All Randomized Subjects Vital Signs Listing 16.2.2.2 All Randomized Subjects Pregnancy Test Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Listing 16.2.2.3 All Randomized Subjects Results Listing 16.2.2.3 All Randomized Subjects Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.2.3 All Randomized Subjects Resement All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.2.5 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.2.6 All Randomized Subjects Surgical Eventocardiogram | Listing 16.2.8.3 | All Randomized Subjects | Non-Medication Therapies |
| Listing 16.2.11 All Randomized Subjects Subject NRS and NRS at Rescue Diary Compliance Listing 16.2.12.1 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.13 All Randomized Subjects Pain Intensity Assessment (NRS with Ambulation) Listing 16.2.13 All Randomized Subjects List of Efficacy Endpoints Listing 16.2.14 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.15 All Randomized Subjects Investigator Global Evaluation (IGE) Listing 16.2.16.1 All Randomized Subjects KOOS - Knee Symptoms Listing 16.2.16.2 All Randomized Subjects KOOS - ADL Listing 16.2.16.3 All Randomized Subjects KOOS - Pain Listing 16.2.16.4 All Randomized Subjects KOOS - Sport/ Rec Listing 16.2.17.1 All Randomized Subjects KOOS - Sport/ Rec Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Serious Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Vital Signs Listing 16.2.19 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.1 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.2 All Randomized Subjects Pregnancy Test Results Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Listing 16.2.2.3 All Randomized Subjects Pregnancy Test Listing 16.2.2.4 All Randomized Subjects Pregnancy Test Listing 16.2.2.5 All Randomized Subjects Roomitation and Targeted Physical Exam Assessment Listing 16.2.2.5 All Randomized Subjects Physical Exam Assessment Listing 16.2.2.5 All Randomized Subjects Pregnancy Test Listing 16.2.2.5 All Randomized Subjects | Listing 16.2.9 | All Randomized Subjects | Surgery |
| Listing 16.2.11. All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.12.1 All Randomized Subjects Pain Intensity Assessment (NRS at Rest) Listing 16.2.13. All Randomized Subjects List of Efficacy Endpoints Listing 16.2.14 All Randomized Subjects List of Efficacy Endpoints Listing 16.2.15 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.16.1 All Randomized Subjects Investigator Global Evaluation (IGE) Listing 16.2.16.2 All Randomized Subjects KOOS - Knee Symptoms Listing 16.2.16.3 All Randomized Subjects KOOS - ADL Listing 16.2.16.4 All Randomized Subjects KOOS - Pain Listing 16.2.16.5 All Randomized Subjects KOOS - Pain Listing 16.2.17.1 All Randomized Subjects KOOS - Quality of Life Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Listing 16.2.18.1 All Randomized Subjects Adverse Events Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Pregnancy Test Listing 16.2.24 All Randomized Subjects Pregnancy Test Listing 16.2.25 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Pregnancy Test Pregnancy Test Listing 16.2.25 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment All Randomized Subjects All Randomized Subjects All Randomized Subjects All Randomize | Listing 16.2.10 | All Randomized Subjects | |
| Listing 16.2.12.1 All Randomized Subjects Listing 16.2.13 All Randomized Subjects Listing 16.2.14 All Randomized Subjects Listing 16.2.15 All Randomized Subjects Listing 16.2.16 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.1 All Randomized Subjects Listing 16.2.16.2 All Randomized Subjects Listing 16.2.16.3 All Randomized Subjects Listing 16.2.16.4 All Randomized Subjects Listing 16.2.16.5 All Randomized Subjects Listing 16.2.17.1 All Randomized Subjects Listing 16.2.17.2 All Randomized Subjects Listing 16.2.17.3 All Randomized Subjects Listing 16.2.17.4 All Randomized Subjects Listing 16.2.18.1 All Randomized Subjects Listing 16.2.18.2 All Randomized Subjects Listing 16.2.18.2 All Randomized Subjects Listing 16.2.18.3 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.18.4 All Randomized Subjects Listing 16.2.2.8 All Randomized Subjects Listing 16.2.2.9 All Randomized Subjects Listing 16.2.22 All Randomized Subjects Listing 16.2.23 All Randomized Subjects Listing 16.2.23 All Randomized Subjects Listing 16.2.24 All Randomized Subjects Listing 16.2.25 All Randomized Subjects Listing 16.2.25 All Randomized Subjects Listing 16.2.25 All Randomized Subjects Listing 16.2.25 All Randomized Subjects Listing 16.2.26 All Randomized Subjects Listing 16.2.27 All Randomized Subjects Listing 16.2.28 All Randomized Subjects Listing 16.2.29 All Randomized Subjects Listing 16.2.20 All Randomized Subjects Listing 16.2.23 All Randomized Subjects Listing 16.2.24 All Randomized Subjects Listing 16.2.25 All Randomized Subjects Listing 16.2.26 All Randomized Subjects Listing 16.2.26 All Randomized Subjects Listing 16.2.26 All Randomized Subjects Listing 16.2.26 All Randomized Subjects Listing 16.2.26 All Randomized Subjects Listing | Listing 16.2.11 | All Randomized Subjects | Subject NRS and NRS at Rescue Diary Compliance |
| Listing 16.2.12.2 All Randomized Subjects List of Efficacy Endpoints Listing 16.2.13 All Randomized Subjects List of Efficacy Endpoints Listing 16.2.14 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.15 All Randomized Subjects Investigator Global Evaluation (IGE) Listing 16.2.16.1 All Randomized Subjects KOOS – Knee Symptoms Listing 16.2.16.2 All Randomized Subjects KOOS – ADL Listing 16.2.16.3 All Randomized Subjects KOOS – Pain Listing 16.2.16.4 All Randomized Subjects KOOS – Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS – Quality of Life Listing 16.2.17.1 All Randomized Subjects Serious Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.1 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Pregnancy Test Listing 16.2.24 All Randomized Subjects Pregnancy Test Listing 16.2.25 All Randomized Subjects Pregnancy Test Listing 16.2.26 All Randomized Subjects Pregnancy Test Listing 16.2.27 All Randomized Subjects Pregnancy Test Listing 16.2.28 All Randomized Subjects Pregnancy Test Listing 16.2.29 All Randomized Subjects Pregnancy Test Listing 16.2.20 All Randomized Subjects Pregnancy Test Listing 16.2.25 All R | | All Randomized Subjects | Pain Intensity Assessment (NRS at Rest) |
| Listing 16.2.14 All Randomized Subjects Patient Global Evaluation (PGE) Listing 16.2.15 | Listing 16.2.12.2 | All Randomized Subjects | Pain Intensity Assessment (NRS with Ambulation) |
| Listing 16.2.14 All Randomized Subjects Investigator Global Evaluation (PGE) Listing 16.2.15 All Randomized Subjects KOOS – Knee Symptoms Listing 16.2.16.2 All Randomized Subjects KOOS – ADL Listing 16.2.16.3 All Randomized Subjects KOOS – ADL Listing 16.2.16.4 All Randomized Subjects KOOS – Pain Listing 16.2.16.5 All Randomized Subjects KOOS – Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS – Quality of Life Listing 16.2.17.1 All Randomized Subjects Serious Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Pregnancy Test Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Pregnancy Test Listing 16.2.24 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam | Listing 16.2.13 | All Randomized Subjects | List of Efficacy Endpoints |
| Listing 16.2.15 All Randomized Subjects KOOS – Knee Symptoms Listing 16.2.16.2 All Randomized Subjects KOOS – ADL Listing 16.2.16.3 All Randomized Subjects KOOS – Pain Listing 16.2.16.4 All Randomized Subjects KOOS – Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS – Quality of Life Listing 16.2.17.1 All Randomized Subjects Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Pregnancy Test Listing 16.2.24 All Randomized Subjects Pregnancy Test Listing 16.2.25 All Randomized Subjects Surgical Examination and Targeted Physical Exam Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam | | All Randomized Subjects | Patient Global Evaluation (PGE) |
| Listing 16.2.16.1 All Randomized Subjects KOOS – Knee Symptoms Listing 16.2.16.2 All Randomized Subjects KOOS – ADL Listing 16.2.16.3 All Randomized Subjects KOOS – Pain Listing 16.2.16.4 All Randomized Subjects KOOS – Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS – Quality of Life Listing 16.2.17.1 All Randomized Subjects Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Examination 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam | | All Randomized Subjects | Investigator Global Evaluation (IGE) |
| Listing 16.2.16.2 All Randomized Subjects KOOS - ADL Listing 16.2.16.3 All Randomized Subjects KOOS - Pain Listing 16.2.16.4 All Randomized Subjects KOOS - Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS - Quality of Life Listing 16.2.17.1 All Randomized Subjects Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Surgical Examination and Targeted Physical Examination 16.2.24 All Randomized Subjects Surgical Site Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam | Y | All Randomized Subjects | KOOS – Knee Symptoms |
| Listing 16.2.16.3 All Randomized Subjects KOOS - Pain Listing 16.2.16.4 All Randomized Subjects KOOS - Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS - Quality of Life Listing 16.2.17.1 All Randomized Subjects Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.29 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Pregnancy Test Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Pregnancy Test Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam | | All Randomized Subjects | KOOS - ADL |
| Listing 16.2.16.4 All Randomized Subjects KOOS – Sport/ Rec Listing 16.2.16.5 All Randomized Subjects KOOS – Quality of Life Listing 16.2.17.1 All Randomized Subjects Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam | | All Randomized Subjects | KOOS - Pain |
| Listing 16.2.16.5 All Randomized Subjects KOOS – Quality of Life Listing 16.2.17.1 All Randomized Subjects Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Examination 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | KOOS – Sport/ Rec |
| Listing 16.2.17.1 All Randomized Subjects Serious Adverse Events Listing 16.2.17.2 All Randomized Subjects Serious Adverse Events Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | |
| Listing 16.2.17.3 All Randomized Subjects Treatment Related Adverse Events Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | _ | All Randomized Subjects | Adverse Events |
| Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | Listing 16.2.17.2 | All Randomized Subjects | Serious Adverse Events |
| Listing 16.2.17.4 All Randomized Subjects Adverse Events Leading to Study Discontinuation Listing 16.2.18.1 All Randomized Subjects Chemistry Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | Treatment Related Adverse Events |
| Listing 16.2.18.1 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.2 All Randomized Subjects Coagulation Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | Adverse Events Leading to Study Discontinuation |
| Listing 16.2.18.2 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.3 All Randomized Subjects Hematology Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | Chemistry Laboratory Test Results |
| Listing 16.2.18.3 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.18.4 All Randomized Subjects Urinalysis Laboratory Test Results Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Examination 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | Coagulation Laboratory Test Results |
| Listing 16.2.18.4 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | All Randomized Subjects | Hematology Laboratory Test Results |
| Listing 16.2.19 All Randomized Subjects Vital Signs Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | Ÿ | All Randomized Subjects | Urinalysis Laboratory Test Results |
| Listing 16.2.20 All Randomized Subjects Alcohol Breath and Urine Drug Screen Tests Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Examination and Targe | <u> </u> | All Randomized Subjects | Vital Signs |
| Listing 16.2.21 All Randomized Subjects Pregnancy Test Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | = | _ |
| Listing 16.2.22 All Randomized Subjects Physical Examination and Targeted Physical Exam Assessment Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | - | |
| Assessment Listing 16.2.23 All Randomized Subjects Knee X-Ray Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | - | |
| Listing 16.2.24 All Randomized Subjects Surgical Site Assessment and Rebound Pain Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | | | |
| Assessment Listing 16.2.25 All Randomized Subjects Neurosensory Exam Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | Listing 16.2.23 | All Randomized Subjects | Knee X-Ray |
| Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | Listing 16.2.24 | All Randomized Subjects | |
| Listing 16.2.26 All Randomized Subjects 12-Lead Electrocardiogram | Listing 16.2.25 | All Randomized Subjects | Neurosensory Exam |
| · | | - | |
| Library 10.2.2. [ 1 17 operation [ 1 harmdookindto (1 17) dondont duton but | Listing 16.2.27 | PK Population | Pharmacokinetic (PK) Concentration Data |


# **14. DOCUMENT HISTORY**

| Version<br># | Summary of Changes | Section Changed | Date |
|---|---|---|---|
| 1.0 | Initial document released | NA | 13MAR2019 |
| 2.0 | Updated for the final protocol version and date. | Various | 24Apr19 |




# **Certificate Of Completion**

Envelope Id: 9FDD589BB9DE4B858939D5ABD00D067E

Subject: Please DocuSign: CA-PS-203 SAP\_Final\_v2.0 24APR2019.pdf

Source Envelope:

Document Pages: 33 Signatures: 3
Certificate Pages: 4 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Enabled

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Status: Completed

**Envelope Originator:** 

Caitlyn Avila

100 W California Blvd., Unit 25

Pasadena, CA 91105 cavila@lotuscr.com

IP Address: 205.197.253.177

#### **Record Tracking**

Status: Original

4/29/2019 2:10:02 PM

Holder: Caitlyn Avila

cavila@lotuscr.com

Location: DocuSign

#### **Signer Events**

Jennifer Nezzer inezzer@lotuscr.com

5:28

Lotus Clinical Research, LLC-Sub Account

Security Level: Email, Account Authentication

(Required)

# Signature

Jennifer Neyyer

Signature Adoption: Pre-selected Style

Signature ID:

F51546CD-923C-410C-87CA-B1F62D450C79

Using IP Address: 45.18.125.80

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I have reviewed this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 8/16/2017 8:46:58 AM

ID: a2e3d9e3-0ef1-4b5e-8f0a-26d3d9799cc6

Mike Royal

Mike@concentricanalgesics.com

Concentric Analgesics, Inc

Security Level: Email, Account Authentication

(Required)

Mike Royal

Signature Adoption: Pre-selected Style

Signature ID:

608C20EC-5FAD-4832-ADC7-99E971759505

Using IP Address: 71.70.192.139

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 5/30/2018 1:05:32 PM

ID: 41453062-babe-431e-8e37-146f718ab8aa

## **Timestamp**

Sent: 4/29/2019 2:12:55 PM Viewed: 4/30/2019 1:21:59 PM Signed: 4/30/2019 1:22:10 PM

Sent: 4/29/2019 2:12:56 PM Viewed: 5/1/2019 7:42:24 AM Signed: 5/1/2019 7:43:06 AM

| Signer Events | Signature | Timestamp |
|---|---|---|
| Song Liou | C 1: | Sent: 4/29/2019 2:12:56 PM |
| sliou@lotuscr.com | Song Liou | Viewed: 4/29/2019 3:37:00 PM |
| Lotus Clinical Research | | Signed: 4/29/2019 3:37:27 PM |
| Security Level: Email, Account Authentication (Required) | Signature Adoption: Pre-selected Style<br>Signature ID:<br>85C80776-CFA1-404F-B9C3-4B43BB0AA100<br>Using IP Address: 108.51.237.84 | |
| | With Signing Authentication via DocuSign passwor | d |
| | With Signing Reasons (on each tab): | |
| | I am the author of this document | |
| Electronic Record and Signature Disclosure: | | |

# Electronic Record and Signature Disclosure: Accepted: 2/16/2018 10:40:34 AM ID: 33003533-520a-46d0-b1ac-311cccf15c53

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 4/29/2019 2:12:56 PM<br>5/1/2019 7:42:24 AM<br>5/1/2019 7:43:06 AM<br>5/1/2019 7:43:06 AM |
| Payment Events | Status | Timestamps |

# ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

Please read the information below carefully and thoroughly. By checking the "I agree to use Electronic Records and Signatures" box in the DocuSign system, you confirm you can access this information electronically to your satisfaction and agree to these terms and conditions below.

# **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after signing session. If you wish for us to send you paper copies of any such documents from our office to you, please contact your Lotus Lead Project Manager.

# Withdrawing your consent

If you decide to receive documents from us electronically, you may at any time change your mind and tell us thereafter that you want to receive documents only in paper format. If you want to withdraw your consent and receive future documents in paper format, please contact your Lotus Lead Project Manager.

# Consequences of changing your mind

If you elect to receive documents only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the documents to you in paper format, and then wait until we receive back from you and your execution of such paper documents. To indicate to us that you are changing your mind within the DocuSign system, you must withdraw your consent using the DocuSign "Withdraw Consent" form on the signing page of a DocuSign envelope instead of signing it. This will indicate to us that you have withdrawn your consent to receive documents electronically from us and you will no longer be able to use the DocuSign system to receive documents electronically from us or to sign electronically documents from us.

# All documents will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all documents that require your signature during the course of our relationship with you. All documents will be sent to you through your e-mail as recorded in the study-specific Study Contact Sheet. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# How to contact Lotus Clinical Research, LLC:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically:

# To advise Lotus Clinical Research, LLC of your new e-mail address

To let us know of a change in your e-mail address, you must send an email message to your Lotus Lead Project Manager and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.

In addition, you must notify DocuSign, Inc. to arrange for your new email address to be reflected

in your DocuSign account by following the process for changing e-mail in the DocuSign system.

# To request paper copies from Lotus Clinical Research, LLC

To request delivery from us of paper copies of the documents previously provided by us to you electronically, you must send an e-mail to your Lotus Lead Project Manager and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number.

# To withdraw your consent

To inform us that you no longer want to receive future documents in electronic format via DocuSign you may:

i. decline to sign a document from within your DocuSign session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send an email to your Lotus Lead Project Manager withdrawing consent, and in the body of such request you must state your e-mail, full name, US Postal Address, and telephone number.

Required hardware and software

| Required hard ware and software | |
|---|---|
| Operating Systems: | Windows® 2000, Windows® XP, Windows |
| | Vista® Mac OS® X |
| Browsers: | Final release versions of Internet Explorer® 6.0 |
| | or above (Windows only); Mozilla Firefox 2.0 |
| | or above (Windows and Mac); Safari <sup>TM</sup> 3.0 or |
| | above (Mac only) |
| PDF Reader: | Acrobat® or similar software may be required |
| | to view and print PDF files |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | Allow per session cookies |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, you will be asked to re-accept the disclosure. Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

# Acknowledging your access and consent to receive materials electronically

By checking the "I agree to use Electronic Records and Signatures" box in the DocuSign system, you are confirming to us that:

- You can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC CONSUMER DISCLOSURES document; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify Lotus Clinical Research, LLC, as described above, you consent to receive through electronic means documents that require your signature